CLINICAL TRIAL: NCT07259980
Title: An Observational Registry-Based Study to Evaluate the Long-Term Safety of Tofersen in People With SOD1-ALS
Brief Title: A Study to Learn More About the Long-Term Safety of Tofersen (Qalsody) in Participants With Superoxide Dismutase 1 (SOD-1) Amyotrophic Lateral Sclerosis (ALS)
Status: Not yet recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 233AS401
Record Dates: First submitted 2025-10-31; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tofersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tofersen: Data for participants with SOD1-ALS will be collected via ALS disease registries, the Treatment Research Initiative to Cure ALS (TRICALS) network's Precision-ALS programme and ALS/MND NHC.
  Interventions: Drug: Tofersen

INTERVENTIONS:
Drug: Tofersen — Administered as specified in the treatment arm.
  Other Names: BIIB067, Qalsody

SUMMARY:
In this study, researchers will learn more about the safety of tofersen, also known as Qalsody®. This is a drug available for doctors to prescribe for participant with a certain type of amyotrophic lateral sclerosis, also known as ALS. This type is in participant who have a mutation in the superoxide dismutase 1 gene, also known as SOD-1.

This is known as an "observational" study, which collects health information about study participants without changing their medical care. Participants for this study will be found using 2 different groups of study research centers that help provide clinical care for participant with ALS. These groups are in Europe and the United States and are called:

* the Precision-ALS programme
* the ALS/Motor Neuron Disease (MND) Natural History Consortium (NHC)

The main goal of this study is to collect safety information in participants with SOD-1 ALS who were in either of the groups.

The main question researchers want to answer in this study is:

* What are the characteristics of the participants in this study?
* How many participants had serious adverse events (SAEs), including ones that affect the brain, spinal cord, or nerves?

An adverse event is a health problem that may or may not be caused by a drug during the study. An adverse event is considered serious when it results in death, is life-threatening, causes lasting problems, or requires hospital care.

Researchers will also learn more about:

* How many participants develop other health conditions or become pregnant, including how the pregnancy turned out
* Why and when participants stopped treatment

This study will be done as follows:

* Participants will be screened to check if they can join the study.
* Data from the participants' regular visits to their clinic will be collected based on which study research center they are in.
* Each participant will be in the study until they decide to leave or until death. Currently, the study is planned to last at least 7 years.

DETAILED DESCRIPTION:
The primary objectives of this study are to describe demographic and clinical characteristics of participants with superoxide dismutase 1-amyotropic lateral sclerosis (SOD1-ALS); to describe the frequency of SAEs among participants with SOD1-ALS, including serious neurologic events previously reported in clinical trial participants (e.g., myelitis, radiculitis, aseptic meningitis, increased intracranial pressure, and/or papilloedema).

The secondary objectives of this study are to describe the frequency of new comorbid conditions, pregnancy and pregnancy outcome among participants with SOD1-ALS; to describe the frequency of treatment discontinuation among participants with SOD1-ALS treated with tofersen.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with an ALS diagnosis and a confirmed SOD1 mutation from contributing registry networks will be considered for inclusion in the study.

Key Exclusion Criteria:

* Data collected while a person with SOD1-ALS is participating in an interventional clinical trial (with tofersen or any other investigational medicinal product) will be excluded.

NOTE: Other protocol- defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with SOD1-ALS enrolled in TRICALS network's Precision-ALS programme with data from participating clinical centers across multiple European countries or at ALS/MND NHC with data from participating clinical centers in the United States (tofersen users and tofersen non-users).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2033-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
Baseline Demographic: Age | At Baseline
Baseline Demographic: Participant Sex | At Baseline
Baseline Demographic: Race/Ethnicity | At Baseline
Baseline Demographic: Weight | At Baseline
Baseline Demographic: Height | At Baseline
Baseline Demographic: Body Mass Index (BMI) | At Baseline
Baseline Demographic: Family History of Amyotrophic Lateral Sclerosis (ALS) | At Baseline
Clinical Characteristics: Age at Diagnosis and Symptom Onset | At Baseline
Clinical Characteristics: Revised El Escorial Classification | At Baseline
Clinical Characteristics: Classification of SOD1-ALS Clinical Phenotypes | At Baseline
Clinical Characteristics: SOD1 Mutation Type | At Baseline
Clinical Characteristics: Medical History | At Baseline
Clinical Characteristics: Concomitant Medications | At Baseline
Clinical Characteristics: Disease History | At Baseline
Clinical Characteristics: Pregnancy Status | At Baseline
Number of Participants With Serious Adverse Events | Up to 7 years

SECONDARY OUTCOMES:
Number of Participants With New Comorbid Conditions | Up to 7 years
Number of Participants With Pregnancy and Pregnancy Outcomes | Up to 7 years
Number of Participants With Reported Treatment Discontinuation | Up to 7 years
Number of Participants With Reported Reasons for Treatment Discontinuation | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org